CLINICAL TRIAL: NCT01907945
Title: Healthy Networks Water Treatment Study
Acronym: HNWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Organic Health Response (Other); Microclinic International (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HNWT
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Household Water Treatment; Waterborne Illness
Keywords: Household water treatment; Waterborne illness; ceramic filters; social network

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participant households in this arm are eligible for participation in the social network-based water treatment education program (referred to as the Microclinic Water Program). Participant households who do not enroll in the Microclinic Water Program receive household-based education identical to that of the 'comparison' arm.
  Interventions: Behavioral: Microclinic Water Program
- Comparison (Active Comparator): Participant households in this arm receive household drinking water treatment education at the household level.
  Interventions: Behavioral: Household education

INTERVENTIONS:
Behavioral: Microclinic Water Program — Three session educational program is delivered to study participants and their self-selected social networks in a group setting. The three session topics are the spread of water borne illness, water treatment methods and social support for sustaining household water treatment. Sessions are taught by a trained community health worker and a study staff member.
  Arms: Intervention
Behavioral: Household education — Three session educational program is delivered to study participants at an individual household level. The three session topics are the spread of water borne illness, water treatment methods and social support for sustaining household water treatment. Sessions are taught by a trained community health worker and a study staff member.
  Arms: Comparison

SUMMARY:
This study is a non-randomized double cohort study evaluating the impact of social network-based water treatment education on sustained household water treatment behaviors over 12 months of follow up. A three-session curriculum was developed on the spread of water borne illness, water treatment methods, and the role of social support in water treatment. Participants in the intervention arm will receive this curriculum in a group setting, where group members are self-selected members of the study participants' social networks. Participants in the comparison arm will receive the same curriculum taught at the individual household level. All participants will receive CeraMaji ceramic filters for use in household water treatment after participating in the three sessions. Research staff will conduct surveys and water quality testing over a period of 12 months to determine whether participants continue to use the ceramic filters. Investigators hypothesize that social network-based training on household water treatment will result in a higher proportion of households using ceramic filters at 6- and 12-months as compared to households receiving individual training.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Mfangano Island Healthy Networks Impact Study
* Resident of Mfangano Island in the East or North sub-locations
* 18 years of age or older
* Conversant in DhoLuo or English

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Ceramic filter use | 6 months post-intervention
  'use' defined as 1) self-reported use in the three days prior to the survey, 2) presence of filter in household and 3) presence of water/moisture in the filter indicating recent use
Ceramic filter use | 12 months post-intervention
  'use' defined as 1) self-reported use in the three days prior to the survey, 2) presence of filter in household and 3) presence of water/moisture in the filter indicating recent use

SECONDARY OUTCOMES:
Fecal coliforms | 6 months post-intervention
  fecal coliforms will be measured in drinking water stored in participant households using the IDEXX QuantiTray 2000 system.
Fecal coliforms | 12 months post-intervention
  fecal coliforms will be measured in drinking water stored in participant households using the IDEXX QuantiTray 2000 system.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Elizabeth Bukusi, MBChB, M.Med, Principal Investigator — Kenya Medical Research Institute; Matthew D Hickey, MD Candidate, Principal Investigator — University of California, San Francisco; Charles R Salmen, MSc, MD candidate, Principal Investigator — University of California, San Francisco
Locations (1):
- Ekialo Kiona Center, Kitawi Beach, Mfangano Island, Nyanza, Kenya

REFERENCES:
- See also: Organic Health Response HNWT page — http://organichealthresponse.org/research/healthy-networks-water-treatment-hnwt/